CLINICAL TRIAL: NCT01229930
Title: CIRCCa - A Randomized Double Blind Phase II Trial of Carboplatin-Paclitaxel Plus Cediranib Versus Carboplatin-Paclitaxel Plus Placebo in Metastatic/Recurrent Cervical Cancer
Brief Title: Carboplatin and Paclitaxel With or Without Cediranib Maleate in Treating Patients With Metastatic or Recurrent Cervical Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Glasgow (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000687338; CRUK-C-2009-01; EUDRACT-2009-011542-25; ISRCTN-23516549; EU-21080; ZENECA-CRUK-C-2009-01
Record Dates: First submitted 2010-10-27; First posted 2010-10-28 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2010-10

CONDITIONS: Cervical Cancer
Keywords: cervical adenocarcinoma; cervical adenosquamous cell carcinoma; cervical squamous cell carcinoma; recurrent cervical cancer; stage IVB cervical cancer; stage IVA cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Carboplatin; cediranib; Paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: cediranib maleate
Drug: paclitaxel
Other: laboratory biomarker analysis
Other: pharmacological study
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Cediranib maleate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. It is not yet known whether carboplatin and paclitaxel are more effective when given with or without cediranib maleate in treating patients with cervical cancer that cannot be removed by surgery.

PURPOSE: This randomized phase II trial is studying giving carboplatin and paclitaxel together with cediranib maleate to see how well it works compared with giving carboplatin and paclitaxel together with a placebo in treating patients with metastatic or recurrent cervical cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To provide preliminary evidence regarding whether the addition of cediranib maleate to a combination of carboplatin and paclitaxel will increase the progression-free survival by 50% from 4 to 6 months in patients with metastatic or recurrent, undetectable cervical carcinoma.

Secondary

* To provide estimates of differences in response, survival, toxicity, quality of life, and pharmacodynamic end-points between the study arms.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive carboplatin IV over 30-60 minutes and paclitaxel IV over 3 hours on day 1. Patients also receive oral placebo once daily.
* Arm II: Patients receive carboplatin and paclitaxel therapy as in Arm I. Patients also receive oral cediranib maleate once daily.

In both arms, treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with complete response, partial response, or stable disease following completion of therapy receive cediranib maleate or placebo until evidence of progression or toxicity.

Blood samples may be collected periodically for evaluation of the VEGFR signaling inhibitor cediranib maleate and identification of suitable biomarkers that predict cediranib maleate response. Quality-of-life is assessed by the EORTC QLQ-C30 and QLQ-CX24 cervix subscale questionnaires at baseline and periodically during study and follow up.

After completion of study therapy, patients are followed up every 2 months for 3 years, every 6 months for 2 years, and then annually thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed carcinoma of the cervix, including any of the following subtypes:

  * Squamous cell carcinoma
  * Adenocarcinoma
  * Adenosquamous cell carcinoma
* Must meet one of the following criteria:

  * Persistent or relapsed inoperable disease after radical radiotherapy within the irradiated pelvis
  * Relapse after radical hysterectomy (after radical radiotherapy to pelvis, if appropriate)
  * Extra pelvic metastases
  * Primary stage IVB disease
* Not suitable for potentially curative surgical procedure
* Measurable disease in ≥ 1 marker site
* No CNS disease, including brain metastases, within the past 6 months

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy > 12 weeks
* Hemoglobin ≥ 10 g/dL
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Calculated creatinine clearance ≥ 35 mL/min
* No proteinuria > 1+ on dipstick (on 2 consecutive dipsticks not less than 1 week apart), unless urinary protein is < 1.5 g in a 24-hour period
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT or AST ≤ 2.5 times ULN (≤ 5 times ULN if hepatic metastases present)
* Alkaline phosphatase ≤ 2.5 times ULN (≤ 5 times ULN if hepatic metastases present)
* Prothrombin ratio (PTR)/INR ≤ 1.5 OR PTR/INR 2.0-3.0 for patients on stable dose of anticoagulant
* Partial thromboplastin time < 1.2 times control
* No history of a nervous or psychiatric disorder that would prevent informed consent and compliance
* No prior malignancy within the past 5 years, except for successfully treated basal cell skin cancer or in-situ breast cancer
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study treatment
* No uncontrolled infection, defined as infection that cannot be resolved readily with antibiotics prior to trial entry
* No history of significant gastrointestinal impairment, as judged by the Investigator, that would significantly affect the absorption of cediranib maleate
* No history of pelvic fistula
* No history of inflammatory bowel disease
* No sub-acute or acute intestinal obstruction
* No significant traumatic injury within the past 4 weeks
* No non-healing wound, ulcer, or bone fracture
* No active bleeding
* No history or evidence of thrombotic or hemorrhagic disorders
* No uncontrolled seizures, cerebrovascular accident, transient ischemic attack, or subarachnoid hemorrhage within the past 6 months
* No significant cardiovascular disease, including any of the following:

  * Arterial thrombotic event within the past 12 months
  * Angina within the past 6 months
  * History of poorly controlled or uncontrolled hypertension or resting BP > 150/100 mm Hg in the presence or absence of a stable regimen of anti-hypertensive therapy within the past 6 months
  * NYHA class II-IV congestive heart failure
  * Peripheral vascular disease ≥ grade 3 or cardiac arrhythmia requiring medication
  * Prolonged QTc (corrected) interval of > 470 ms on ECG or a family history of long QT syndrome
* Patients with rate-controlled atrial fibrillation are eligible
* Not requiring intravenous nutritional support
* No preexisting sensory or motor neuropathy ≥ grade 2
* No history or clinical suspicion of spinal cord compression
* No known hypersensitivity to carboplatin or paclitaxel
* No evidence of any other disease, metabolic dysfunction, physical examination finding, or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No unresolved toxicity ≥ CTC grade 2 from prior systemic anti-cancer therapy, except hematological toxicity or alopecia
* No prior chemotherapy, except cisplatin administered along with radiotherapy as primary treatment
* No major surgery within 28 days or anticipated while on study
* More than 2 weeks since prior and no concurrent potent inhibitors of CYP3A4 and 2C8, including any of the following:

  * Amiodarone
  * Clarithromycin
  * Erythromycin
  * Simvastatin
  * Atorvastatin
  * Lovastatin
  * Montelukast sodium
  * Verapamil
  * Ketoconazole
  * Miconazole
  * Indinavir (and other antivirals)
  * Diltiazem
* No concurrent grapefruit juice or St. John wort

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Overall progression-free survival

SECONDARY OUTCOMES:
Reduction in plasma VEGFR2 levels from baseline to day 28
Response to chemotherapy using RECIST1.1 criteria
Overall survival
Toxicity assessed using NCI CTCAE v4.0
Quality of life assessed using EORTC QLQ-C30 and CX24

CONTACTS AND LOCATIONS:
Overall Officials: R. Paul Symonds, MD, FRCP, FRCR, Principal Investigator — University Hospitals, Leicester
Locations (5):
- United Kingdom (5):
  - Leicester Royal Infirmary, Leicester, England
  - Cancer Research UK and University College London Cancer Trials Centre, London, England
  - Christie Hospital, Manchester, England
  - Royal Marsden - Surrey, Sutton, England
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland